CLINICAL TRIAL: NCT03182725
Title: Effect of Ivabradine on Patients With Postural Orthostatic Tachycardia Syndrome (a Double-blind Placebo-parallel Group Trial)
Brief Title: Effect of Ivabradine on Patients With Postural Orthostatic Tachycardia Syndrome
Acronym: POTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Pam Taub, MD, Associate Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 170694
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: POTS; tachycardia; ivabradine
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Tachycardia | interventions — Ivabradine

STUDY DESIGN:
Intervention Model Description: 20 patients with POTS will receive Ivabradine treatment vs placebo for one month. Then there will be a one-month wash out period prior to the cross over in which patients who received Ivabradine will receive the placebo, and patients who initially were on placebo will now receive Ivabradine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patient will consume one placebo pill twice a day for one month.
  Interventions: Drug: Placebo
- Ivabradine (Experimental): Patient will consume one dose of Ivabradine twice a day for one month.
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — Ivabradine is prescribed for treatment of chronic heart failure through inhibition of the f-channels (If) within the sinoatrial node.
  Arms: Ivabradine
Drug: Placebo — A substance that has no therapeutic effect and will act as a control.
  Arms: Placebo

SUMMARY:
Postural orthostatic tachycardia syndrome (POTS) occurs in approximately 500,000 Americans, but predominates in women with a 5:1 ratio. Patients with POTS experience debilitating tachycardia upon postural changes such as standing that impairs their quality of life. Tachycardia is clinically defined as a heart rate greater than 100 beats/min; and in POTS patients, the prolonged heart rate increase is greater than 30 beats/min or increases to 120 beats/min within the first ten minutes of a diagnostic tilt table test without postural hypotension. There are currently no effective treatment methods for POTS. However, several studies suggest Ivabradine could be a main treatment option for POTS because Ivabradine specifically inhibits the f-channels (If) within the sinoatrial (SA) node, which slows the heart rate. Currently in the US, Ivabradine is mainly prescribed to treat chronic heart failure. It is well tolerated in patients, but it is not commonly prescribed for POTS. It has been also used for treatment of inappropriate sinus tachycardia with good benefit. The hypothesis for this experiment is that Ivabradine will reduce tachycardia and improve functional status in patients with POTS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-65.
* Subjects must have POTS diagnosis (Hyperadrenergic Subtype with NE> 600pg/ml))
* Subjects with no structural heart disease
* Subject with no arrhythmias
* Subjects with norepinephrine levels greater than 600 pg/ml
* Subjects with normal CBC, Metabolic, and thyroid levels

Exclusion Criteria:

* Thyroid or adrenal disorders
* Drugs that interfere with Ivabradine (example: Cytochrome P450 drugs)
* Presentation of peripheral edema and discolored toes with peripheral autonomic neuropathy. Symptoms include: legs (reduced hair growth, cramps), toes (blue color), legs/feet (wounds, ulcers that do not heal), and muscles (numbness, heaviness)
* Subjects who have had a history of systemic illnesses (acute or chronic infectious); autoimmune/ inflammatory disease, cancer, COPD, anemia, diabetes, or psychiatric illness
* Subjects with resting heart rate< 60beats/min, atrial fibrillation, advanced AV blocks, sinus disease, and acute decompensated heart failure and severe hepatic impairment.
* Smokers or alcohol abuse
* Pregnant or breastfeeding mothers
* Woman of childbearing potential who are unwilling to use highly effective contraception during treatment and for an additional one month after discontinuing the study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pam Taub, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Result] McDonald C, Frith J, Newton JL. Single centre experience of ivabradine in postural orthostatic tachycardia syndrome. Europace. 2011 Mar;13(3):427-30. doi: 10.1093/europace/euq390. Epub 2010 Nov 9. PMID 21062792
- [Result] Ewan V, Norton M, Newton JL. Symptom improvement in postural orthostatic tachycardia syndrome with the sinus node blocker ivabradine. Europace. 2007 Dec;9(12):1202. doi: 10.1093/europace/eum235. Epub 2007 Oct 19. No abstract available. PMID 17951266
- [Result] Barzilai M, Jacob G. The Effect of Ivabradine on the Heart Rate and Sympathovagal Balance in Postural Tachycardia Syndrome Patients. Rambam Maimonides Med J. 2015 Jul 30;6(3):e0028. doi: 10.5041/RMMJ.10213. PMID 26241226

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 participants signed the consent form but did not pass the screening assessments. 1 participant signed the consent form and then withdrew prior to randomization.
Groups:
- Placebo in Arm A, Ivabradine in Arm B: In the first Arm, Patient will consume one placebo pill twice a day for one month. After the first arm, there will be a one-week washout. After washout, the patient will commence Arm B where they consume ne dose of ivabradine twice a day for one month.
  Placebo: A substance that has no therapeutic effect and will act as a control.
  In the second arm, patient will consume one dose of Ivabradine twice a day for one month.
  Ivabradine: Ivabradine is prescribed for treatment of chronic heart failure through inhibition of the f-channels (If) within the sinoatrial node.
- Ivabradine in Arm A, Placebo in Arm B: Patient will consume one dose of Ivabradine twice a day for one month. In the first Arm, Patient will consume one dose of ivabradine twice a day for one month. After the first arm, there will be a one-week washout. After washout, the patient will commence Arm B where they consume one placebo pill twice a day for one month
  Placebo: A substance that has no therapeutic effect and will act as a control.
  In the second arm, patient will consume one dose of Ivabradine twice a day for one month.
  Ivabradine: Ivabradine is prescribed for treatment of chronic heart failure through inhibition of the f-channels (If) within the sinoatrial node.
Period: Treatment Arm 1 (First Half of Study)
Arm/Group | Placebo in Arm A, Ivabradine in Arm B | Ivabradine in Arm A, Placebo in Arm B
Started | 16 | 10
Completed | 16 | 7
Not Completed | 0 | 3
Period: Treatment Arm 2 (Second Half of Study)
Arm/Group | Placebo in Arm A, Ivabradine in Arm B | Ivabradine in Arm A, Placebo in Arm B
Started | 16 | 6 (One participant withdrew during crossover and therefore did not start Treatment Arm 2.)
Completed | 16 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo in Arm A, Ivabradine in Arm B: In the first Arm, Patient will consume one placebo pill twice a day for one month.
  Placebo: A substance that has no therapeutic effect and will act as a control.
  In the second arm, patient will consume one dose of Ivabradine twice a day for one month.
  Ivabradine: Ivabradine is prescribed for treatment of chronic heart failure through inhibition of the f-channels (If) within the sinoatrial node.
- Ivabradine in Arm A, Placebo in Arm B: In the first arm of the study, patient will consume one dose of Ivabradine twice a day for one month.
  Ivabradine: Ivabradine is prescribed for treatment of chronic heart failure through inhibition of the f-channels (If) within the sinoatrial node.
  In the second arm, patient will consume one placebo pill twice a day for one month.
  Placebo: A substance that has no therapeutic effect and will act as a control.
- Total: Total of all reporting groups
Arm/Group | Placebo in Arm A, Ivabradine in Arm B | Ivabradine in Arm A, Placebo in Arm B | Total
Number analyzed (Participants) | 16 | 10 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 10 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.75 (10.7) | 27.8 (11.15) | 34.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 10 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 10 | 23
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Heart Rate
Description: Orthostatic heart rate monitoring will be used to gauge heart rate changes.
Time Frame: Baseline and one month post-treatment
Population: In total, 22 patients with hyperadrenergic POTS as the predominant subtype completed a randomized, double-blinded, placebo-controlled, crossover trial with ivabradine. Patients were randomized to start either ivabradine or placebo for 1 month, and then were crossed over to the other treatment for 1 month. Heart rate, QOL, and plasma NE levels were measured at baseline and at the end of each treatment month.
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Placebo: In the first Arm, Patient will consume one placebo pill twice a day for one month.
  Placebo: A substance that has no therapeutic effect and will act as a control.
Arm/Group | Placebo | Ivabradine
Number analyzed (Participants) | 22 | 22
beats per minute | 17.0 (10.4) | 13.1 (8.6)

2. Secondary Outcome: Change in Quality of Life Via SF-36 Survey
Description: Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) The SF-36 has 36 questions and is an indicator of overall health status and is well-validated. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. The total score on the SF-36 ranges from 0 - 100 Lower scores = more disability, higher scores = less disability
  Sections:
  Vitality Physical functioning Bodily pain General health perceptions Physical role functioning Emotional role functioning Social role functioning Mental health
Time Frame: Baseline and one month post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ivabradine
Number analyzed (Participants) | 22 | 22
units on a scale | 44.1 (22.4) | 53.4 (27)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events were monitored in all enrolled participants over a period of 3 months.
Arm/Group | Placebo | Ivabradine
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

LIMITATIONS AND CAVEATS:
* smaller sample size
* many patients suspected they were on ivabradine
* patients were only on 1 month of ivabradine; longer study duration may be warranted to assess potential long term effects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT03182725/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT03182725/ICF_001.pdf